CLINICAL TRIAL: NCT00831675
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity Among Healthy Children Receiving Influenza Virus Vaccine Fluzone® 2004-2005
Brief Title: Study of Safety and Immunogenicity of Fluzone® in Healthy Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC21
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2009-08-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® vaccine; Infants; Toddlers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infants <12 Months (Experimental): Participants aged ≥ 6 to < 12 months at enrollment and received 2 doses of Fluzone® Vaccine
  Interventions: Biological: Influenza Vaccine 2004-2005 Paediatric Formulation
- Toddlers ≥12 Months (Experimental): Participants aged ≥ 12 to < 36 months at enrollment and received 2 doses of Fluzone® vaccine
  Interventions: Biological: Influenza Vaccine 2004-2005 Paediatric Formulation

INTERVENTIONS:
Biological: Influenza Vaccine 2004-2005 Paediatric Formulation — 0.25 mL (Day 0 and Day 28), Intramuscular
  Other Names: Fluzone®
  Arms: Infants <12 Months
Biological: Influenza Vaccine 2004-2005 Paediatric Formulation — 0.25 mL (Day 0 and Day 28), Intramuscular
  Other Names: Fluzone®
  Arms: Toddlers ≥12 Months

SUMMARY:
To describe the safety of the 2004-2005 pediatric formulation of the inactivated, split-virion influenza vaccine Fluzone®, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months.

To describe the immunogenicity of the 2004-2005 inactivated, split-virion influenza vaccine Fluzone®, administered in a two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to < 36 months

DETAILED DESCRIPTION:
To provide the Centers for Biologic Evaluation and Research (CBER) with sera collected from healthy children receiving the 2004-2005 formulation of the inactivated, split-virion influenza vaccine Fluzone® for further study by the Food and Drug Administration (FDA), Centers for Disease Control and Prevention (CDC), and the World Health Organization (WHO).

ELIGIBILITY:
Inclusion Criteria :

* Participant is aged ≥ 6 months to < 36 months.
* Participant is considered to be in good health on the basis of reported medical history and limited physical examination.
* Participant is available for the duration of the study.
* Parent/guardian is willing and able to provide informed consent.
* Parent/guardian is willing and able to meet protocol requirements.

Exclusion Criteria :

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* Previous history of influenza vaccination or documented history of influenza infection.
* An acute illness with or without fever (temperature > 100.4 °F rectal) in the 72 hours preceding enrollment in the trial (defer enrollment).
* Clinically significant findings in vital signs or review of systems (investigator judgment; defer or exclude).
* Participation in any other clinical trial within 30 days prior to enrollment up to termination of the subject's participation in the study.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known human immunodeficiency virus (HIV)-positive mother.
* Prior history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 3.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants took part in the study from 16 September through 18 November 2004 in 1 US site.
Pre-assignment Details: A total of 30 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Infants <12 Months: Participants aged ≥ 6 to < 12 months at enrollment and received 0.25 mL intramuscular injection of Fluzone® vaccine on Day 0 and on Day 28, respectively.
- Toddlers ≥12 Months: Participants aged ≥ 12 to < 36 months at enrollment and received 0.25 mL intramuscular injection of Fluzone® vaccine on Day 0 and on Day 28, respectively.
Period: Overall Study
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Started | 12 | 18
Completed | 12 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants <12 Months | Toddlers ≥12 Months | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 18 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 8.9 (2.1) | 20 (6.0) | 15.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Reactions After Vaccination With Fluzone® 2004-2005 Pediatric Formulation
Description: Solicited local reactions: Erythema, bruising, induration, pain at injection site.
  Solicited systemic reactions: Fever (temperature), irritability, crying, lethargy, appetite decreased, diarrhea, vomiting, rash collected daily for four days after each injection.
Time Frame: Days 0-3 Post-dose
Population: Safety analysis was on all enrolled and vaccinated subjects with available reaction data, intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Number analyzed (Participants) | 12 | 18
Participants
  Any Solicited Local Reaction Post-dose 1 | 3 | 7
  Any Erythema (>0.5 cm) | 0 | 2
  Grade 3 Erythema (>5.0 cm) | 0 | 0
  Any Induration (>0.5 cm) | 0 | 0
  Grade 3 Induration (>5.0 cm) | 0 | 0
  Any Bruising (>0.5 cm) | 0 | 0
  Grade 3 Bruising (>5.0 cm) | 0 | 0
  Any Pain | 3 | 5
  Grade 3 Pain (Cry When inj. Limb is Moved) | 0 | 0
  Any Solicited Local Reaction Post-dose 2 | 4 | 4
  Any Erythema (> 0.5 cm) | 2 | 0
  Grade 3 Erythema (>5.0 cm) | 0 | 0
  Any Induration (>0.5 cm) | 0 | 0
  Grade 3 Induration (>5.0 cm) | 0 | 0
  Any Bruising (>0.5 cm) | 2 | 0
  Grade 3 Bruising (>5.0 cm) | 0 | 0
  Any Pain | 4 | 4
  Grade 3 Pain (Cry When inj. Limb Is Moved) | 0 | 0
  Any Solicited Systemic Reaction Post-dose 1 | 7 | 12
  Any Fever | 0 | 3
  Grade 3 Fever (>103.1 ºF) | 0 | 0
  Any Irritability | 5 | 9
  Grade 3 Irritability (>3 hours) | 0 | 1
  Any Crying | 3 | 6
  Grade 3 Crying (>3 hours) | 0 | 0
  Any Lethargy | 1 | 1
  Grade 3 Lethargy (Disabling) | 0 | 0
  Any Appetite Decreased | 1 | 4
  Grade 3 Appetite Decreased (refuses over 3 feeds) | 0 | 0
  Any Vomiting | 1 | 1
  Grade 3 Vomiting (3 or more episodes) | 0 | 1
  Any Diarrhea | 3 | 1
  Grade 3 Diarrhea (>5 Diarrhea Stools) | 0 | 0
  Rash - Presence of Welts | 1 | 1
  Any Solicited Systemic Reaction Post-dose 2 | 6 | 10
  Any Fever | 1 | 3
  Grade 3 Fever (>103.1 ºF) | 0 | 0
  Any Irritability | 5 | 6
  Grade 3 Irritability (>3 hours) | 1 | 0
  Any Crying | 4 | 3
  Grade 3 Crying (>3 hours) | 0 | 0
  Any Lethargy | 1 | 1
  Grade 3 Lethargy (Disabling) | 0 | 0
  Any Appetite Decreased | 3 | 6
  Grade 3 Appetite Decreased (refuses 3 feeds) | 0 | 0
  Any Vomiting | 1 | 2
  Grade 3 Vomiting (3 or more episodes) | 0 | 0
  Any Diarrhea | 3 | 0
  Grade 3 Diarrhea (>5 Diarrhea Stools) | 0 | 0
  Rash - Presence of Welts | 1 | 0

2. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Antibodies Pre- and Post-Vaccination With Fluzone® Vaccine 2004-2005 Pediatric Formulation
Time Frame: 14 days post-vaccination
Population: GMTs were evaluated in the per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Number analyzed (Participants) | 12 | 18
Titers
  A/New Caledonia/20/99, Pre-dose | 7.9 [6.4 to 9.9] | 9.4 [7.0 to 12.8]
  A/New Caledonia/20/99, Post-dose | 15.0 [11.2 to 20.1] | 26.2 [15.8 to 43.3]
  A/Wyoming/03/2003, Pre-dose | 7.9 [4.8 to 13.2] | 14.4 [6.5 to 31.8]
  A/Wyoming/03/2003, Post-dose | 31.7 [12.9 to 78.2] | 108.9 [44.8 to 264.7]
  B/Jiangsu/10/2003, Pre-dose | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  B/Jiangsu/10/2003, Post-dose | 7.5 [5.0 to 11.1] | 8.4 [6.5 to 10.8]

3. Other Pre Specified Outcome: Percentage of Participants With at Least a 40 Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination (Seroprotection)
Description: Seroprotection defined as percentage of participants with reciprocal hemagglutination inhibition titers ≥40 post-vaccination with Fluzone®.
Time Frame: 14 days post-vaccination
Population: Seroprotection were evaluated in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Number analyzed (Participants) | 12 | 18
Percentage of Participants
  A/New Caledonia/20/99 | 8 | 39
  A/Wyoming/03/2003 | 50 | 67
  B/Jiangsu/10/2003 | 8 | 0

4. Other Pre Specified Outcome: Percentage of Participants With a 4-Fold Increase in Serum Hemagglutination Inhibition Antibody Titers Post-Vaccination (Seroconversion)
Description: Seroconversion defined as the percentage of participants with a ≥ 4-fold increases in titer from pre- to post-vaccination with Fluzone®.
Time Frame: Day 14 post-vaccination
Population: Seroconversion were evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Number analyzed (Participants) | 12 | 18
Percentage of Participants
  A/New Caledonia/20/99 | 33 | 50
  A/Wyoming/03/2003 | 58 | 100
  B/Jiangsu/10/2003 | 8 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of vaccination to Day 42 post-vaccination.
Arm/Group | Infants <12 Months | Toddlers ≥12 Months
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 11/12 | 14/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants <12 Months (N=12) | Toddlers ≥12 Months (N=18)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea NOS (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 7 (9) | 3 (3)
Vomiting NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 4 (4)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis NOS (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media NOS (Infections and infestations) | 3 (3) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis NOS (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection NOS (Infections and infestations) | 5 (5) | 2 (2)
Upper respiratory tract infection viral NOS (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
Dermatitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications